CLINICAL TRIAL: NCT07036315
Title: An Investigation of the Intersection of Affect and Meaning in Music-Based Pain Modulation
Brief Title: Meaning in Music-Based Pain Modulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Patrick Finan, PhD, Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSR 230193; U24AT012601 (NIH)
Record Dates: First submitted 2025-06-13; First posted 2025-06-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: The Focus of the Study is Healthy Volunteers
Keywords: Music; Pain; Meaning
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain-Modulation (Experimental): Participants will be exposed to different music clips.
  Interventions: Other: Music intervention

INTERVENTIONS:
Other: Music intervention — Participants will be asked to select different music clips based on meaning, enjoyment and preference.

SUMMARY:
The overall goal of this project is to examine the impact of music's meaning on pain. Relationships between trait affect, meaning in life, and subjective qualities of meaningful music will be assessed. We will also conduct interviews with a subset of participants to determine which aspects of music are most meaningful and how this meaning increases or decreases pain sensations.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Absence of acute or chronic pain
* Normal hearing (either naturally or with assistance of hearing device)
* Must be able to wear an EEG
* Able to sign consent

Exclusion Criteria:

* < 18 or > 65 years old
* Presence of acute pain (brief pain inventory score > 3)
* Pregnant women
* Participant reports that they experience pain on more days than not in the past 6 months (i.e., chronic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Pain Unpleasantness | Baseline/Pre-intervention and During the Intervention
  Participants will be asked to report pain unpleasantness on a 1 - 100 visual analogue scale ranging from 0 (no sensation) to 100 (intolerable pain)
Pain Intensity | Baseline/Pre-intervention and During the Intervention
  Participants will be asked to report pain intensity on a 1 - 100 visual analogue scale ranging from 0 (no sensation) to 100 (intolerable pain)

SECONDARY OUTCOMES:
The Multidimensional Meaning in Life Scale | Baseline/Pre-intervention
  The multidimensional meaning in life scale is a 16 item validated questionnaire that measures judgments about life's meaning including three subscales of coherence, purpose and mattering. Participants respond to each item using a 7-point Likert scale (1 = Very strongly disagree, 7 = Very strongly agree). A higher score indicates a stronger sense of that dimension of meaning in life.
The Positive and Negative Affect Schedule-X (PANAS-X) | Baseline/Pre-Intervention
  The Positive and Negative Affect Schedule-X (PANAS-X) is a 60-item measure assessing perceived intensity of various emotions, which are aggregated to form positive and negative affect scales, and a series of subscales. Scores are calculated by summing the numerical values of a 5-point Likert type scale (1 = Very slightly or not at all, 5 = extremely) for each item. Higher scores indicate higher levels of the specific affect being measured.
The Hedonic and Eudaimonic Motives for Activities Scale | Baseline/Pre-intervention
  The Hedonic and Eudaimonic Motives for Activities scale is a 9 item survey used to assess how participants typically approach activities in daily life. Participants rate each item on a 7-point Likert type scale (1 = not at all, 7 = very much) with higher scores indicating more hedonic or eudaimonic motives for activities.
The Geneva Emotional Music Scale | During the Intervention
  Participants will be asked to rate their affective responses to each music clip on a 9-point Likert-type scale. Higher scores indicate a greater experience of each emotion measured.
Optional Micro-Phenomenological Interview | Immediately After the Intervention
  The objective of the interview is to gain in-depth data on participants' thoughts and feelings about what makes music meaningful to them and how such meaning relates to their experience of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No